CLINICAL TRIAL: NCT03503812
Title: Mitigating the Health Effects of Desert Dust Storms Using Exposure-Reduction Approaches: Assessment of Health Outcomes in Children With Asthma and in Adults With Atrial Fibrillation During Desert Dust Storms (With vs Without Interventions)
Brief Title: Mitigating the Health Effects of Desert Dust Storms Using Exposure-Reduction Approaches
Acronym: MEDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Collaborators: University of Crete (Other); Soroka University Medical Center (Other); Cyprus University of Technology (Other); Department of Labor Inspection, Ministry of Labor, Welfare and Social Insurance, Cyprus (Unknown); Department of Meteorology, Ministry of Agriculture, Rural Development and Environment, Cyprus (Unknown); Cyprus Broadcasting Corporation (Unknown); E.n.A Consulting LP (Unknown)
Responsible Party: Principal Investigator, Panayiotis Yiallouros, Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LIFE MEDEA Protocol
Record Dates: First submitted 2018-03-22; First posted 2018-04-20 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Asthma in Children; Atrial Fibrillation
Keywords: Randomized clinical trial; Public Health Intervention; Behavioral Intervention; Exposure-Reduction Approaches; Desert dust storm events; Climate change; Asthma in children; Atrial Fibrillation; Air pollution
MeSH Terms: conditions — Atrial Fibrillation | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Following the eligibility assessment, we will randomize each group of participants (group with asthmatic children and group with AF patients) with a 1:1:1 ratio to three parallel groups to receive: a) no intervention for DDS, b) intervention for outdoor exposure reduction, by reducing the time spend outdoors and by avoiding physical activity, c) interventions for outdoor (as above) and indoor exposure reduction (by minimizing home ventilation and filtering indoor air). In the indoor intervention arm of the study, exposure reduction measures will be applied in the asthmatic child's classroom/school and bedroom/household settings and in the AF patient's household/bedroom settings. The study design offers also the opportunity to assess: 1.outdoor exposures to PM, and 2.indoor exposures to PM and related health outcomes in three parallel groups during the same DDS events with and without intervention measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No intervention to DDS exposure - Asthma in Children (No Intervention)
- Intervention 1 - Asthma in Children (Experimental)
  Interventions: Behavioral: Intervention (1) for outdoor exposure reduction - Asthma in Children
- Intervention 2 - Asthma in Children (Experimental)
  Interventions: Behavioral: Intervention (2) for outdoor and indoor exposure reduction - Asthma in Children
- No intervention to DDS exposure - Atrial Fibrillation (No Intervention)
- Intervention 1 - Atrial Fibrillation (Experimental)
  Interventions: Behavioral: Intervention (1) for outdoor exposure reduction - Atrial Fibrillation
- Intervention 2 - Atrial Fibrillation (Experimental)
  Interventions: Behavioral: Intervention (2) for outdoor and indoor exposure reduction - Atrial Fibrillation

INTERVENTIONS:
Behavioral: Intervention (1) for outdoor exposure reduction - Asthma in Children — Intervention 1 (I1) aims to reduce exposure to outdoor particles and it will be applied on days with DDS during the follow-up period. This intervention will consist of two recommendations:
  1. Reduce time spent outdoors and
  2. Reduce physical activity
  Arms: Intervention 1 - Asthma in Children
Behavioral: Intervention (2) for outdoor and indoor exposure reduction - Asthma in Children — Intervention 2 (I2) aims to reduce both:
  i) exposure to outdoor particles and it will be applied on days with DDS during the follow-up period. This intervention will consist of two recommendations:
  1. Reduce time spent outdoors and
  2. Reduce physical activity
     ii) indoor particle levels on a continuous daily basis throughout the follow-up DDS period. This intervention will consist of two recommendations for participants' schools and houses:
  3. Reduce particle infiltration into residences by keeping windows and doors closed as much as possible and
  4. Reduce indoor particle levels by using air cleaners.
  Arms: Intervention 2 - Asthma in Children
Behavioral: Intervention (1) for outdoor exposure reduction - Atrial Fibrillation — Intervention 1 (I1) aims to reduce exposure to outdoor particles and it will be applied on days with DDS during the follow-up period. This intervention will consist of two recommendations:
  1. Reduce time spent outdoors and
  2. Reduce physical activity
  Arms: Intervention 1 - Atrial Fibrillation
Behavioral: Intervention (2) for outdoor and indoor exposure reduction - Atrial Fibrillation — Intervention 2 (I2) aims to reduce both:
  i) exposure to outdoor particles and it will be applied on days with DDS during the follow-up period. This intervention will consist of two recommendations:
  1. Reduce time spent outdoors and
  2. Reduce physical activity
     ii) indoor particle levels on a continuous daily basis throughout the follow-up DDS period. This intervention will consist of two recommendations for participants' houses:
  3. Reduce particle infiltration into residences by keeping windows and doors closed as much as possible and
  4. Reduce indoor particle levels by using air cleaners.
  Arms: Intervention 2 - Atrial Fibrillation

SUMMARY:
The MEDEA project is envisioned to provide the field-based evidence for the adoption of a strategic plan for mitigating the health effects of desert dust storm (DDS) events in South-Eastern Europe. Over the past decade, several studies have demonstrated that DDS in Mediterranean countries, originating mostly from the Sahara and Arabian Peninsula deserts, have been increasing in number and magnitude and linked it to desertification, climatic variability and global warming. EU legislation considers DDS impossible to prevent, implicitly harmless and discounts their contribution to daily and annual air quality standards of particulate matter up to 10 microns (PM10). However, there is increasing evidence from epidemiological studies, which correlates exposure to PM10 during DDS with a significant increase in mortality and hospital admissions from cardiovascular and respiratory causes. Therefore, there is a pressing need for EU policies to reduce population exposures and increase individual, population and institutional resilience to the growing frequency and intensity of DDS. MEDEA ultimate goal is to demonstrate the feasibility and effectiveness of an adaptation strategy to DDS and better inform EU policy making. The adaptation strategy will be carried out within two panel studies, with two different groups of patients; 1. Children with asthma and 2. Adults with atrial fibrillation (AF). The primary objective will be to quantify the vulnerability of children with asthma and adults with AF during DDS outbreaks and provide evidence-based estimates demonstrating which interventions/recommendations work best in mitigating adverse health effects in this group of patients after randomization of each group of patients to three parallel intervention groups: a) No intervention for DDS; b) Intervention for outdoor exposure reduction, and c) Interventions for both outdoor and indoor exposure reduction. The secondary objective of the study is to demonstrate which of the recommendations are effective in reducing outdoor and indoor exposures to DDS in a panel of children with asthma and in a panel of AF adults.

Intervention: Each group of patients (children with asthma and AF patients) will be recruited and will be randomized during the high DDS outbreaks season (Spring 2019 and 2020) with 1:1:1 ratio into three parallel groups to receive: a) No intervention for DDS; b) Intervention for outdoor exposure reduction, by reducing the time spend outdoors and by avoiding physical activity and c) Interventions for outdoor (as above) and indoor exposure reduction (by minimizing home ventilation and filtering indoor air). Disease-related adverse health outcomes will be assessed in the three parallel arms of the study.

Approaches for delivering the intervention: A bidirectional, patient-centered e-Platform will be developed in order to facilitate prompt communication with the participants and provide early warnings regarding forecasted upcoming DDS events through text messaging and smartphone applications. Furthermore, the same IT platform and mobile application will be utilised for the dissemination of the exposure reduction guidelines that the participants will follow.

Assessment of adherence to intervention: 1.Monitor compliance to exposure-reduction guidelines using remote sensors. The intervention for outdoor exposure reduction, entailing reduction of the time spend outdoors and avoidance of physical activity, will be assessed with the use of smart wristwatches that will be equipped with Global Positioning System (GPS) and an accelerometer. 2.The intervention for indoor exposure reduction, entailing minimization of home ventilation and filtering of indoor air, will be assessed with the use of particle samplers that will be placed outside and inside of houses and school classrooms.

DETAILED DESCRIPTION:
Study design for the panel study with asthmatic children:

Children with asthma will be recruited during DDS outbreaks and will be randomized into three parallel groups to receive:

1. No intervention for DDS,
2. Intervention for outdoor exposure reduction, and
3. Interventions for both outdoor and indoor exposure reduction.

Disease-related adverse health outcomes will be assessed in all the parallel arms of the study.

Previous publications of the MEDEA investigators, indicated that 2/3 of each year's DDS events in the Eastern Mediterranean region appear during February-May, with 10-15% of the days during this period being "DDS days". Thus, the investigators will perform this panel study during February-May of 2019, and 2021. In addition, the panel study will run in September - December (a period also characterized with frequent DDS events) of the same years.

Study population, sample size and location: Children with mild to moderate persistent asthma, aged 6-11 years, will be recruited from primary schools in Nicosia-Cyprus (n=150) in academic years 2018-2019, 2019-2020 and 2020-2021. In order to facilitate recruitment, schools principals will be contacted individually at the beginning of each academic year and details of the study will be explained. Relations with the Administrative and Nursing staff of the Schools and Parents Associations will be established with the aim to facilitate field work. During fall 2018, 2019 and 2021, MEDEA investigators will start recruitment efforts to detect eligible children with asthma for participation in the study in the high DDS periods of February-May 2019 and 2020. The same number of children will be recruited at the second study site of Heraklion-Crete.

With an average number of 250 students per school, a childhood asthma prevalence of 9-10% and an estimated response of 60%, in 18-20 primary schools we expect to detect 300 students with reported asthma. We expect that 50% of the children with reported asthma will meet eligibility criteria giving us for randomization 150 subjects in Nicosia. We estimate a dropout rate of 30%, which will eventually give us 105 asthmatic children in total to analyze.

The feasibility of protocols to assess health outcomes with and without implementation of exposure reduction guidelines will be tested in a pilot study during the high DDS outbreaks season of 2018 at both study sites in a small number of patients (6 children with asthma per study site).

Duration of the study: A feasibility trial and refinement of protocols and tools will be performed in the high DDS period of 2018 (February-May). In fall 2018 and 2019, with the onset of academic year, screening survey questionnaires (International Study of Asthma and Allergies in Children, ISAAC) will be addressed to the parents of all children in 18-20 primary schools in Nicosia by the MEDEA investigators to detect eligible asthmatic children for participation in the study during the upcoming high DDS periods of February-May 2019 and 2020.

Study Enrollment Procedures: Children with mild to moderate persistent asthma, aged 6-11 years, will be recruited at primary schools in Nicosia-Cyprus (n=150) in academic years 2018-2019, 2019-2020 and 2020-2021. In order to facilitate recruitment, schools' principals will be contacted individually at the beginning of each academic year and details of the study will be explained. Relations with the Administrative and Nursing staff of the Schools and Parents Associations will be established with the aim to facilitate field work. With the use of screening questionnaires (ISAAC questionnaires), parents will, after giving written consent, report their child's respiratory health information. Then the parents of children with asthmatic symptoms will be invited to participate in the MEDEA program after they give their written consent. For children participating in the program, consent to their participation will be given by their parents/guardians. Parents will be asked by the study investigators to read the respective consent forms for the survey and the study, and will be given the opportunity to ask any clarification questions for their child's participation.

Interventions, Administration, and Duration: Following the eligibility assessment, we will randomize participating schools (and their students with asthma) with a 1:1:1 ratio to three parallel groups to receive:

1. no intervention for DDS
2. intervention for outdoor exposure reduction, by reducing the time spend outdoors and by avoiding physical activity
3. interventions for outdoor (as above) and indoor exposure reduction (by minimizing home ventilation and filtering indoor air).

In the indoor intervention arm of the study, exposure reduction measures will be applied in the asthmatic child's classroom/school and bedroom/household settings.

After randomization, the children, their parents and schoolteachers will be trained in the tools and procedures to be followed.

Prior to the high DDS season, each eligible child will have at the school:

* baseline demographic, medical, and symptom survey, and
* assessments of lung function (Spirometry), fractional exhaled nitric oxide (FeNO), and specific aero-allergen sensitivities.

The study design offers also the opportunity to assess:

* outdoor exposures to PM,
* indoor exposures to PM and
* related health outcomes in three parallel groups during the same DDS events with and without intervention measures

Handling of Study Interventions:

A bidirectional, patient-centered e-Platform will be created to:

* Communicate promptly forecast alerts to individuals about upcoming DDS events through smartphone applications and text messaging
* Disseminate exposure reduction guidelines

In particular, in the group where there will be intervention for outdoor exposure reduction, the intervention will be carried out by:

* Informing the participant and the parent for upcoming desert dust storm episodes.
* Simultaneous transmission of instructions to a smartphone to reduce outdoor exposure during the episode (stay indoors, avoid intense physical activity outdoors, avoid competitive sports, avoid unnecessary walks).

In the group where there will be interventions for outdoor and indoor exposure reduction, the intervention will be carried out by:

* Informing the participant and the parent for upcoming desert dust storm episodes.
* Simultaneous transmission of instructions to a smartphone to reduce:

  1. Outdoor exposure during the episode (stay indoors, avoid intense physical activity outdoors, avoid competitive sports, avoid unnecessary walks) and
  2. Indoor, home and classroom exposure (closed windows and doors, sealing possible cracks around windows and doors in order to minimize home ventilation, and using an air cleaner in order to filter indoor air).

Adherence Assessment: The compliance to exposure-reduction guidelines will be monitored with the use of remote sensors. The intervention for outdoor exposure reduction, (by reducing the time spend outdoors and by avoiding physical activity) will be assessed with the use of smart wristwatches that will be equipped with Global Positioning System (GPS) and accelerometer. The intervention for indoor exposure reduction (by minimizing home ventilation and by filtering indoor air) will be assessed with the use of particle samplers that will be placed outside and inside of houses and school classrooms.

Assessment of adverse events: Since, the intervention under study is behavioral/lifestyle intervention, it does not involve any specific drug administration nor any change in ongoing medication regimen. Furthermore, it does not include any invasive procedure and all the health outcomes are assessed using non-invasive methods (smart-watches, phone interviews) and questionnaires. Hence, there are no specific safety parameters to quantify adverse health events related to interventions.

At any point during the study, patients will have the opportunity to bring any information or issue (e.g. health issue) that concerns them to the attention of the primary investigator, whose contact information will be given to all participants during the enrollment phase, and will also be available on the program's website.

Intervention discontinuation:Subjects may withdraw voluntarily from the study at any time and for any reason.

Parents or guardians of asthmatic children can make oral complaints to members of the research team as well as to the principal investigators of each site.

The criteria for discontinuation of intervention will be:

* Non-adherence to the intervention
* Moving to a different house than the reported initial one
* Moving to a different school
* Significant change in health status

Study design for the panel study with the AF patients:

Patients with AF will be recruited during DDS outbreaks and will be randomized into three parallel groups to receive:

1. No intervention for DDS,
2. Intervention for outdoor exposure reduction, and
3. Interventions for both outdoor and indoor exposure reduction.

Disease-related adverse health outcomes will be assessed in all the parallel arms of the study.

Previous publications of the MEDEA investigators, indicated that 2/3 of each year's DDS events in the Eastern Mediterranean region appear during February-May, with 10-15% of the days during this period being "DDS days". Thus, the investigators will perform this public health intervention study during February-May of 2019 and 2020. In addition, the panel study will run in September - December (a period also characterized with frequent DDS events) of the same years.

Study population, sample size and location: Men and women with prior implantation of a dual lead (atrial and ventricular) pacemaker or implantable cardioverter defibrillator (ICD), will be recruited from cardiac arrhythmia clinics in General Hospital in Nicosia-Cyprus (n=156) in project years 2018-2019, 2019-2020 and 2020-2021. Recruitment of participants will be facilitated through the network of physicians in Nicosia General Hospital. In order to facilitate recruitment, relations will be established with the Administrative and Nursing staff of the Clinics and Patients' Associations and the details of the project will be explained to them. During fall 2018, 2019, 2020 and 2021, MEDEA investigators will start recruitment efforts to detect eligible AF patients for participation in the study in the high DDS periods of February-May and September-December of 2019, 2021 and 2022.

The same number of patients will be recruited in each study site (Beer Sheba, Heraklion, Nicosia) and the investigators expect that a total of 468 AF patients will be recruited. The investigators estimate a dropout rate of 30%, which will eventually give 324 AF patients to analyse. The feasibility of protocols to assess health outcomes in vulnerable patient groups will be tested in the pilot study during the high DDS outbreaks season of 2018 with and without implementation of exposure reduction guidelines in all study sites in a small number of patients (6 AF patients per study site).

Duration of the study: A feasibility trial and refinement of protocols and tools will be performed in the high DDS period of 2018 (February-May). In the fall of 2018, 2019,2020, 2021 and 2022, MEDEA investigators will start recruitment efforts to detect eligible AF patients for participation in the study during the high DDS periods of February-May and September-December 2019, 2020, 2021 and 2022.

Study Enrolment Procedures: Men and women with prior implantation of a dual lead (atrial and ventricular) pacemaker or ICD, will be recruited from the cardiac arrhythmia clinic at Nicosia General Hospital in Cyprus (n=156) in project years 2018-2019, 2019-2020, 2020-2021 and 2021-2022. Recruitment of participants will be facilitated through the network of physicians at Nicosia General Hospital. In order to facilitate recruitment, relations will be established with the Administrative and Nursing staff of the Clinic and Patients' Association and the details of the project will be explained to them. Patients will be able to ask questions and ask for clarification on all aspects of the program. Each patient participating in the program should complete the necessary consent forms.

Interventions, Administration, and Duration: Following recruitment, the investigators will randomize participants with a 1:1:1 ratio to three parallel groups to receive:

1. no intervention for DDS
2. intervention for outdoor exposure reduction, by reducing the time spend outdoors and by avoiding physical activity
3. interventions for outdoor (as above) and indoor exposure reduction (by minimizing home ventilation and filtering indoor air).

In the indoor intervention arm of the study, exposure reduction measures will be applied in the patient's household/bedroom settings.

After randomization, and prior to the high DDS season, each eligible participant will complete a questionnaire, providing socio-demographic characteristics, detailed medical and medication history, and will be trained in the tools and procedures to be followed during the monitoring sessions while in the community.

The study design offers also the opportunity to assess:

* outdoor exposures to PM,
* indoor exposures to PM and
* related health outcomes in three parallel groups during the same DDS events with and without intervention measures

Handling of Study Interventions: A bidirectional, patient-centered e-Platform will be created to:

* Communicate promptly forecast alerts to individuals about upcoming DDS events through smartphone applications and text messaging
* Disseminate exposure reduction guidelines

In particular, in the group where there will be intervention for outdoor exposure reduction, the intervention will be carried out by:

* Informing the participant for upcoming desert dust storm episodes.
* Simultaneous transmission of instructions to patient's smartphone to reduce outdoor exposure during the episode (stay indoors, avoid intense physical activity outdoors, avoid competitive sports, avoid unnecessary walks).

In the group where there will be interventions for outdoor and indoor exposure reduction, the intervention will be carried out by:

* Informing the participant for upcoming desert dust storm episodes.
* Simultaneous transmission of instructions to patient's smartphone to reduce a) outdoor exposure during the episode (stay indoors, avoid intense physical activity outdoors, avoid competitive sports, avoid unnecessary walks), and b) indoor, home exposure (closed windows and doors, sealing possible cracks around windows and doors in order to minimize home ventilation, and using an air cleaner in order to filter indoor air).

Adherence Assessment: The compliance to exposure-reduction guidelines will be monitored with the use of remote sensors. The intervention for outdoor exposure reduction, (by reducing the time spend outdoors and by avoiding physical activity) will be assessed with the use of smart wristwatches that will have global position system (GPS) and accelerometer. The intervention for indoor exposure reduction (by minimizing home ventilation and by filtering indoor air) will be assessed with the use of particle samplers that will be placed outside and inside houses.

Assessments of adverse events: Since, the intervention under study is behavioral/lifestyle intervention, it does not involve any specific drug administration nor any change in ongoing medication schedule. Furthermore, it does not include any invasive procedure and all the health outcomes are assessed using non-invasive methods (smart-watches, phone interviews) and questionnaires. Hence, there are no specific safety parameters to quantify adverse health events related to interventions.

At any point during the study, patients will have the opportunity to bring any evolving information or issue (e.g. health issue) that concerns them to the attention of the primary investigator, whose contact information will be given to all participants during the enrollment phase, and will also be available on the program's website.

Intervention discontinuation: Subjects may withdraw voluntarily from the study at any time and for any reason.

Patients can make oral complaints to members of the research team as well as to the principal investigators of each site.

The criteria for intervention discontinuation will be:

* Non-adherence to the intervention
* Moving to a different house than the reported initial one
* Significant change in health status

ELIGIBILITY:
Inclusion Criteria for Children with asthma:

The inclusion criteria for this panel study will be children with physician-diagnosed asthma for at least one year and with at least one of the following:

* Anti-asthma medication in the past year,
* Wheezing in the past year, or
* An unscheduled medical visit for asthma in the past year.

Exclusion Criteria for Children with asthma:

The exclusion criteria will be:

* Lung disease other than asthma
* Cardiovascular disease
* Not living at least 5 days per week in the household

Inclusion Criteria for AF patients:

The inclusion criteria for this panel study will be patients with permanent dual lead (atrial and ventricular) pacemaker or ICD implanted at least two months prior to randomization, with:

* A history of AF or
* Detection of AF in pacemaker/ICD monitoring

Exclusion Criteria for AF patients:

The exclusion criteria will be:

* Permanent AF
* Patients with reversible causes of AF (eg hyperthyroidism)
* Inability to understand and use study tools (smartphones, software applications)
* Terminal illness
* Active smoking
* Not living at least 5 days per week in the household.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Asthma Control Test (ACT) questionnaire score between the no intervention group and the intervention groups in asthmatic children during the high DDS period of 2019 | 4 months
  An improvement of more than 3 points in the ACT or an ACT score>=20 during the high DDS period will be considered. The ACT is a 5-item patient-based assessment that measures dimensions of asthma control. Each item is assessed on a 5-point scale. The scores are summed to give a total score ranging from 5-25. A score of>=20 denotes 'well-controlled asthma', a score of 16-19 denotes 'not well-controlled asthma', and a score of<=15 denotes 'very poorly controlled asthma'. Each month, the combined effect of the ACT will be compared in the two intervention groups vs. the no intervention group. Next, investigators will compare between each of the intervention groups and no intervention group and between the intervention groups. A validated-Greek ACT will be performed via phone interviews at baseline and then at every 1 month during the high DDS period. The frequency of respiratory symptoms will be assessed via child's responses to questions on daytime-night-time symptoms in the past 4 weeks
Comparison of Asthma Control Test (ACT) questionnaire score between the no intervention group and the intervention groups in asthmatic children during the high DDS period of 2020 | 4 months
  An improvement of more than 3 points in the ACT or an ACT score>=20 during the high DDS period will be considered. The ACT is a 5-item patient-based assessment that measures dimensions of asthma control. Each item is assessed on a 5-point scale. The scores are summed to give a total score ranging from 5-25. A score of>=20 denotes 'well-controlled asthma', a score of 16-19 denotes 'not well-controlled asthma', and a score of<=15 denotes 'very poorly controlled asthma'. Each month, the combined effect of the ACT will be compared in the two intervention groups vs. the no intervention group. Next, investigators will compare between each of the intervention groups and no intervention group and between the intervention groups. A validated-Greek ACT will be performed via phone interviews at baseline and then at every 1 month during the high DDS period. The frequency of respiratory symptoms will be assessed via child's responses to questions on daytime-night-time symptoms in the past 4 weeks
Comparison of the number and duration of high atrial frequency episode between the no intervention group and the intervention groups in adults with AF during the high DDS period of 2019. | 6 months
  AF burden is defined as the overall time percentage with AF during the observed period. An AF episode is considered every detected high atrial frequency episode of >330 ms (180 beats per minute) lasting for longer than 30 s with an atrial sensitivity of 0.5 mV. For the primary analysis, the investigators will compare the combined effect in the two intervention groups versus the no intervention (control) group. Secondarily, the effectiveness of each intervention will be compared versus the no intervention (control group) and to each other.
Comparison of the number and duration of high atrial frequency episode between the no intervention group and the intervention groups in adults with AF during the high DDS period of 2020. | 6 months
  AF burden is defined as the overall time percentage with AF during the observed period. An AF episode is considered every detected high atrial frequency episode of >330 ms (180 beats per minute) lasting for longer than 30 s with an atrial sensitivity of 0.5 mV. For the primary analysis, the investigators will compare the combined effect in the two intervention groups versus the no intervention (control) group. Secondarily, the effectiveness of each intervention will be compared versus the no intervention (control group) and to each other.

SECONDARY OUTCOMES:
Comparison of the secondary outcome measures between the no intervention group and the 2 intervention groups during the high DDS period of 2019 | 4 months
  Secondary outcome measures: presence or absence of asthma symptoms in the prior 4-week period, asthma medication use, unscheduled visits for asthma, forced expiratory volume in 1 second, peak expiratory flow, and FeNO
Comparison of the secondary outcome measures between the no intervention group and the 2 intervention groups during the high DDS period of 2020 | 4 months
  Secondary outcome measures: presence or absence of asthma symptoms in the prior 4-week period, asthma medication use, unscheduled visits for asthma, forced expiratory volume in 1 second, peak expiratory flow, and FeNO
Comparison of secondary outcome measures between the no intervention group and the intervention groups in adults with AF during the high DDS period of 2019. | 6 months
  Secondary outcome measures: occurrence of the ventricular arrythmias (assessed through the pacemaker) and heart rate variability
Comparison of secondary outcome measures between the no intervention group and the intervention groups in adults with AF during the high DDS period of 2020. | 6 months
  Secondary outcome measures: occurrence of the ventricular arrythmias (assessed through the pacemaker) and heart rate variability
Comparison of air pollution exposure between the no intervention group and the two intervention groups in children with Asthma during the high DDS periods | 4 months
  Exposure to levels of PM2.5 and PM10 (assessed through particle cascade impactors and particle optical sensors)
Comparison of air pollution exposure between the no intervention group and the two intervention groups in adults with AF during the high DDS periods | 6 months
  Exposure to levels of PM2.5 and PM10 (assessed through particle cascade impactors and particle optical sensors)
Comparison of health related quality of life between the no intervention group and the two intervention groups in adults with AF during the high DDS periods | 6 months
  Changes in Atrial Fibrillation Effect on Quality of life survey (AFEQT questionnaire)
Comparison of arrhythmia medication use between the no intervention group and the two intervention groups in adults with AF during the high DDS periods | 6 months
  Changes in arrhythmia medication
Comparison of unscheduled hospital visits between the no intervention group and the two intervention groups in adults with AF during the high DDS periods | 6 months
  Changes in unscheduled hospital visits

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Yiallouros, MD, PhD, Principal Investigator — Medical School, University of Cyprus
Locations (3):
- Medical School, University of Cyprus, Nicosia, Aglantzia, Cyprus
- School of Medicine, University of Crete, Heraklion, Crete, Greece
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Achilleos S, Evans JS, Yiallouros PK, Kleanthous S, Schwartz J, Koutrakis P. PM10 concentration levels at an urban and background site in Cyprus: the impact of urban sources and dust storms. J Air Waste Manag Assoc. 2014 Dec;64(12):1352-60. doi: 10.1080/10962247.2014.923061. PMID 25562931
- [Background] Gerasopoulos E, et al. Origin and variability of particulate matter (PM10) mass concentrations over the Eastern Mediterranean. Atmos Environ 2006; 40:4679-4690.
- [Background] Griffin DW. Atmospheric movement of microorganisms in clouds of desert dust and implications for human health. Clin Microbiol Rev. 2007 Jul;20(3):459-77, table of contents. doi: 10.1128/CMR.00039-06. PMID 17630335
- [Background] Krasnov H, Katra I, Koutrakis P, Friger MD. Contribution of dust storms to PM10 levels in an urban arid environment. J Air Waste Manag Assoc. 2014 Jan;64(1):89-94. doi: 10.1080/10962247.2013.841599. PMID 24620406
- [Background] Leski TA, Malanoski AP, Gregory MJ, Lin B, Stenger DA. Application of a broad-range resequencing array for detection of pathogens in desert dust samples from Kuwait and Iraq. Appl Environ Microbiol. 2011 Jul;77(13):4285-92. doi: 10.1128/AEM.00021-11. Epub 2011 May 13. PMID 21571877
- [Background] Mallone S, Stafoggia M, Faustini A, Gobbi GP, Marconi A, Forastiere F. Saharan dust and associations between particulate matter and daily mortality in Rome, Italy. Environ Health Perspect. 2011 Oct;119(10):1409-14. doi: 10.1289/ehp.1003026. PMID 21970945
- [Background] Middleton N, Yiallouros P, Kleanthous S, Kolokotroni O, Schwartz J, Dockery DW, Demokritou P, Koutrakis P. A 10-year time-series analysis of respiratory and cardiovascular morbidity in Nicosia, Cyprus: the effect of short-term changes in air pollution and dust storms. Environ Health. 2008 Jul 22;7:39. doi: 10.1186/1476-069X-7-39. PMID 18647382
- [Background] Neophytou AM, Yiallouros P, Coull BA, Kleanthous S, Pavlou P, Pashiardis S, Dockery DW, Koutrakis P, Laden F. Particulate matter concentrations during desert dust outbreaks and daily mortality in Nicosia, Cyprus. J Expo Sci Environ Epidemiol. 2013 May-Jun;23(3):275-80. doi: 10.1038/jes.2013.10. Epub 2013 Feb 20. PMID 23423218
- [Background] Querol X, et al. African dust contributions to mean ambient PM10 mass-levels across the Mediterranean, Basin. Atmos Environ 2009; 43:4266-4277
- [Background] Samoli E, Nastos PT, Paliatsos AG, Katsouyanni K, Priftis KN. Acute effects of air pollution on pediatric asthma exacerbation: evidence of association and effect modification. Environ Res. 2011 Apr;111(3):418-24. doi: 10.1016/j.envres.2011.01.014. PMID 21296347
- [Background] Vodonos A, et al. The impact of desert dust exposures on hospitalizations due to exacerbation of chronic obstructive pulmonary disease. Air Qual Atmos Health 2014; 7:433-439
- [Derived] Kouis P, Galanakis E, Michaelidou E, Kinni P, Michanikou A, Pitsios C, Perez J, Achilleos S, Middleton N, Anagnostopoulou P, Dimitriou H, Revvas E, Stamatelatos G, Zacharatos H, Savvides C, Vasiliadou E, Kalivitis N, Chrysanthou A, Tymvios F, Papatheodorou SI, Koutrakis P, Yiallouros PK. Improved childhood asthma control after exposure reduction interventions for desert dust and anthropogenic air pollution: the MEDEA randomised controlled trial. Thorax. 2024 May 20;79(6):495-507. doi: 10.1136/thorax-2023-220877. PMID 38388489
- [Derived] Anagnostopoulou P, Kouis P, Papatheodorou SI, Middleton N, Papasavvas I, Avraamides P, Simantirakis E, Anastasiou I, Novack V, Stamatelatos G, Revvas E, Kaniklides C, Tymvios F, Savvides C, Koutrakis P, Yiallouros PK. MEDEA randomised intervention study protocol in Cyprus, Greece and Israel for mitigation of desert dust health effects in adults with atrial fibrillation. BMJ Open. 2023 Mar 24;13(3):e069809. doi: 10.1136/bmjopen-2022-069809. PMID 36963790
- [Derived] Kouis P, Papatheodorou SI, Kakkoura MG, Middleton N, Galanakis E, Michaelidi E, Achilleos S, Mihalopoulos N, Neophytou M, Stamatelatos G, Kaniklides C, Revvas E, Tymvios F, Savvides C, Koutrakis P, Yiallouros PK. The MEDEA childhood asthma study design for mitigation of desert dust health effects: implementation of novel methods for assessment of air pollution exposure and lessons learned. BMC Pediatr. 2021 Jan 6;21(1):13. doi: 10.1186/s12887-020-02472-4. PMID 33407248

DOCUMENTS (3):
  • Study Protocol: MEDEA Protocol for Asthmatic Children (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03503812/Prot_000.pdf
  • Study Protocol: MEDEA Protocol for AF patients (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03503812/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03503812/SAP_002.pdf